CLINICAL TRIAL: NCT04955405
Title: The 7-Visit Transition of Care Hospital to Home Intervention: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Allyson G. Hall, Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 3000006289
Record Dates: First submitted 2021-06-16; First posted 2021-07-08 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Chronic Obstructive Pulmonary Disease; Chronic Heart Failure
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Seven telemedicine visits (Experimental): Will receive the seven visit telemedicine protocol
  Interventions: Other: The seven visit telemedicine protocol
- Control - Usual Care (No Intervention): Will not receive the protocol

INTERVENTIONS:
Other: The seven visit telemedicine protocol — The transition of care team (pharmacist, advanced practice provider, social worker) will conduct an initial visit as a team with the patient using the telemedicine platform. During the visit, the team will assess the clinical, social, and pharmaceutical needs of the patient. The transition of care team will then meet to discuss the specific needs of the patient and to develop a care plan for the next 6 telemedicine visits. Either the social worker or the advanced practice provider will conduct the next 6 visits. The pharmacist will provide medication counseling as needed and recommended by the entire care team. The next 3 visits will occur weekly, the following 2 visits will occur biweekly, and the remaining 1 visit will occur at some point during the third month.
  Arms: Seven telemedicine visits

SUMMARY:
New approaches to care transitions must deploy a longer-term and more intensive program that provide an array of services that address underlying social determinants of health (e.g. lack of adequate social support, lack of self-efficacy in managing symptoms and medications, impoverished living conditions, inability to connect with primary care and access. In addition, programs must be adaptable to meet the specific needs of individual patients. Our collaboration of health services researchers, quantitative scientists, and physicians propose to develop and implement a 90-day intensive and comprehensive intervention to support newly discharged patients with COPD and/or CHF. The proposed intervention will utilize a three-person team (registered nurse, clinical social worker, and a pharmacist) to provide an array of medical and social services specifically targeted to meet the needs of individual patients and their families.

Aim: To determine using a randomized control trial, whether participation in an intensive series of 7 home-visits that provide tailored medical and social services among newly discharged low-income Medicare patients with COPD and/or CHF results in a) better patient-reported outcomes and b) a reduced likelihood of repeat hospital care (ED use or hospitalization) relative to a group of patients who receive usual discharge instructions.

DETAILED DESCRIPTION:
The long-term objective of this study is to inform and enhance the ability of UAB Hospitalist Medicine (UABHM) and UAB Health System (UABHS) reduce the likelihood of unplanned readmissions among discharged patients with a diagnosis of chronic obstructive pulmonary disease (COPD) and/or chronic heart failure (CHF). The project involves the implementation of a series of 7 telemedicine visits over 3 months to 35 patients recently discharged from UAB Hospital Medicine.

The Intervention Prior to discharge from the hospital 70 eligible patients will be recruited by physicians who are a part of the hospital medicine service. Thirty-five patients will be assigned to a treatment group and 35 patients to a control group. Consent will be obtained prior to discharge

Intervention Group: Either prior to discharge or during an initial phone call once they are home, patients will be introduced to the telemedicine technology platform. They will also be asked to complete a baseline survey that asks questions about the care transition process from the hospital to home, informational support, physical function, self-efficacy, and emotional distress. An appointment will be set for the patient's first visit with the care transition intervention team.

During the initial first visit, the advanced practice provider will conduct a medical assessment, the social worker will assess living and psychosocial conditions. The pharmacist

The transition of care team (pharmacist, advanced practice provider, social worker) will conduct an initial visit as a team with the patient using the telemedicine platform. During the visit, the team will assess the clinical, social, and pharmaceutical needs of the patient. The pharmacist will conduct medication reconciliation with a review of the patient's medication profile in totality and cross comparing the medications with all comorbid disease states to assure that no additional medications are warranted at that time. The pharmacist will then run the medications through a number of trusted databases such as Lexicomp or Clinical Pharmacology to confirm that there are no harmful drug-drug interactions that require modification prior to discharge.

The transition of care team will then meet to discuss the specific needs of the patient and to develop a care plan for the next 6 telemedicine visits. Either the social worker or the advanced practice provider will conduct the next 6 visits. The pharmacist will provide medication counseling as needed and recommended by the entire care team. Notes from each telemedicine encounter will be developed and stored in RedCap for team review.

The next 3 visits will occur weekly, the following 2 visits will occur biweekly, and the remaining 1 visit will occur at some point during the third month.

Participants will be asked to complete a baseline survey, and follow-up surveys at the end of the 4th week and again at the end of week 12.

Control Group: The control group will complete a baseline survey, and follow-up surveys at the end of the 4th week and at week 12.

ELIGIBILITY:
Inclusion Criteria:

* English Speaking
* Chronic Heart Failure
* Chronic Obstructive Pulmonary Disease
* Age 60 years and older
* Able to provide consent

Exclusion Criteria:

* Does not provide consent
* Cognitive Impairment
* Less than 60 years
* Non-English Speaking

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2022-01-31 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Hospital revisits (Emergency Department or Inpatient) | 90 days
  A measure of whether a participant returned to the University of Alabama at Birmingham (UAB) Emergency Department or had an inpatient admission to UAB for any cause between 24 hours and 90 days following discharge from an index discharge. This measure will be calculated from UAB Health System Electronic Health record data.
  Bivariate and multivariate comparisons will be made between the intervention and control groups
Self-reported declarations on hospital revisits (Emergency Department or Inpatient) | 90 days
  Participant self-report of any hospital visit or emergency department visit within 90 days following discharge from UAB Hospital
  Bivariate and multivariate comparisons between the intervention and control groups

SECONDARY OUTCOMES:
Self efficacy for managing medication and treatment | baseline (day following discharge), 30 and 90 days (following discharge)
  Patient-reported measure comes from the PROMIS item bank (Self-Efficacy for Managing Medication and Treatment, v1.0 short form available from: https://www.healthmeasures.net/search-view-measures?task=Search.search)
  Calculation of score: Each of 4 items has five response options (1=not at all confident, 2=a little confident; 3=somewhat confident; 4=quite confident; 5=very confident) . Response to each question will be summed into a raw score. Raw scores will range from 20 to 4 The raw score will then located on an applicable conversion table maintained by the PROMIS, to translate the raw score into a T-score for each participant. The T-score rescales the raw score into a standardized score. Higher scores are a better outcome.
  Analysis: Compare self-efficacy between intervention and control groups at 30 and 90 days; Compare the change in self-efficacy between 30 and 90 days between intervention and control groups

OTHER OUTCOMES:
National Quality Forum's 3-item Care Transition Measure | baseline (day following discharge); 30 days (following discharge)
  The 3-item care transition measure rates patient perceptions of information provided at hospital discharge. This will be measured at baseline (within one day of discharge and within 30 days of the discharge from the hospital.
  Response categories for each item range: Strongly Disagree=1; disagree=2; Agree=3; Strong Agree=4. Scores will be summed and divided by total possible score. Will use linear transformation to convert to a 0 to 100 scale. Higher scores represent a better outcome (See National Quality Forum, Specifications for the Three-Item Transition Measure available at: https://mhdo.maine.gov/_pdf/NQF_CTM_3_%20Specs_FINAL.pdf),
  Analysis: Compare intervention and control groups at baseline and at 30 days. Compare the change in score between baseline and 30 days between intervention and control groups

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham Health System, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No